CLINICAL TRIAL: NCT04886375
Title: The Effect of USG- Guided Modified Pectoral Nerve Block and Erector Spinae Plane Block on Postoperative Analgesia in Video Assisted Thoracoscopic Surgery
Brief Title: Comparison of USG- Guided Modified Pectoral Nerve Block and Erector Spinae Plane Block on Postoperative Analgesia in Video Assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Sertçakacılar, MD, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-124
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Analgesia; Video-assisted Thoracoscopic Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esp group (Active Comparator): The investigators performed erector spina plane block to that patient group for postoperative analgesia
  Interventions: Procedure: erector spina plane block
- pecs group (Active Comparator): The investigators performed modified pectoral nerve block to that patient group for postoperative analgesia
  Interventions: Procedure: modified pectoral nerve block

INTERVENTIONS:
Procedure: erector spina plane block — The investigators performed erector spina plane block to that patient group for postoperative analgesia
  Arms: esp group
Procedure: modified pectoral nerve block — The investigators performed modified pectoral block to that patient group for postoperative analgesia
  Arms: pecs group

SUMMARY:
This study aims to compare the effects of the erector spinae plan block (ESP) and modified pectoral nerve block (PECS II) on postoperative analgesia in patients undergoing video- assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
55 patients (ASA I-II-III) between 18 and 65 years of age, who were to undergo VATS, were randomized and divided into two groups. (26 patients in each of the PECS and ESP groups). Three patients were excluded from the study because thoracotomy was performed. ESP block was performed for ESP group and a modified pectoral nerve block was performed in the PECS group. Postoperative analgesia was provided by intravenous morphine infusion using a patient-controlled analgesia device. Postoperative 24-hour total morphine consumption and duration of analgesia were the primary outcome measure. Perioperative remifentanil use, numeric rating scale values, time of the first analgesic request, and additional analgesic consumption were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-65
* Patients who will undergo VATS
* ASA I-II-III patients

Exclusion Criteria:

* Clinically diagnosis of spinal or chest wall deformity or pathology
* Clinically known local anesthetic allergy
* Morbid obesity (body mass index>40 kg m2)
* Clinically diagnosis of opioid, alcohol and substance dependence
* Clinically diagnosis of psychiatric disease
* Coagulopathy
* Patients with ASA IV-V

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative 24-hours total morphine consumption | 24 hours postoperatively
  This will be measured only one time by pca device at the 24th hour after surgery.

SECONDARY OUTCOMES:
NRS scores of patients | 24 hours postoperatively
  NRS at 0, 1, 2, 4, 8, 12 ve 24th hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided